CLINICAL TRIAL: NCT03190317
Title: Health Information for Infected Veterans
Acronym: HI-FIV
Status: Active, not recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IIR 15-327
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: electronic medical record; personal health record; Veteran; self-management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- HIV-infected Veterans who use MHV: This group represents the population of HIV-infected Veterans active in care at a VA health system, who have been diagnosed with HIV and use MHV.
  Interventions: Other: HIV-infected Veterans who use MHV
- HIV-infected Veterans who do not use MHV: This group represents the population of HIV-infected Veterans active in care at a VA health system, who have been diagnosed with HIV and do not use MHV.
  Interventions: Other: HIV-infected Veterans who do not use MHV
- Providers and staff of HIV-infected veteran: This groups represents the population of providers and staff who utilize the MHV portal to deliver care for HIV-infected veterans.
  Interventions: Other: Providers and staff of HIV-infected veteran

INTERVENTIONS:
Other: HIV-infected Veterans who use MHV — The investigators will use information from Veteran medical records to assess the relationship between Veteran HIV health care outcomes and the use of MHV. Next, the investigators will interview Veterans to understand why MHV is used. Finally, the investigators will create an intervention based on the information learned that will encourage use of MHV and ask Veterans to test it out.
  Groups: HIV-infected Veterans who use MHV
Other: HIV-infected Veterans who do not use MHV — The investigators will use information from Veteran medical records to assess the relationship between Veteran HIV health care outcomes and the use of MHV. Next, the investigators will interview Veterans to understand why MHV is not used. Finally, the investigators will create an intervention based on the information learned that will encourage use of MHV and ask Veterans to test it out.
  Groups: HIV-infected Veterans who do not use MHV
Other: Providers and staff of HIV-infected veteran — The investigators will interview providers and staff to understand why they think Veterans at their health system use or do not use the MHV portal for self management. The investigators will create and test an intervention based on information learned that will encourage use of MHV among Veterans and providers/staff.
  Groups: Providers and staff of HIV-infected veteran

SUMMARY:
This is a study of My HealtheVet (MHV) use by Veterans diagnosed with Human Immunodeficiency Virus (HIV) and VA providers/staff who care for them. The investigators hope to learn and understand how MHV can improve the self-management of chronic conditions like HIV. First, the investigators will review Veteran medical records to look at the relationship between use of MHV and whether it has a positive or negative impact on the Veteran's management of HIV. Next, the investigators will interview participants to find out how MHV for self-management is used by Veterans and to find out why Veterans and providers choose to use (or not use) specific MHV tools. Lastly, the investigators will use the information found from the first two steps and create an intervention that will encourage non-MHV users to use the MHV tools that can help achieve health-related goals. Once the intervention has been developed, Veterans and providers will participate in a "cognitive walkthrough" to help the researchers test the intervention to see if it is usable, possible, and acceptable.

DETAILED DESCRIPTION:
Over the last twenty years, HIV has transformed from a terminal disease to a condition with near normal life expectancy for patients who follow ideal treatment regimens. HIV-infected individuals still face many challenges and need to be active in self-management of HIV and other conditions in order to live a healthy life. In order to ensure that this population of HIV-infected individuals actively self-manages the condition, personal health records (PHRs) should be used more often. PHRs may simplify disease self-management, improve health outcomes, and reduce unnecessary health care use.

The VA has one of the nation's largest PHR systems - My HealtheVet (MHV). MHV includes features that can help patient's self-manage the disease (e.g., prescription refill, viewing lab results view, secure messaging). While there has been recognition that MHV holds promise as a self-management tool, there has not yet been an examination of use of MHV features and the relationship to health outcomes in any chronic disease group, let alone in HIV-infected Veterans.

The objective of this project is to evaluate MHV use by HIV-infected Veterans and providers, by completing three aims/steps.

Aim/Step 1: Describe the relationship between use of MHV tools for self-management across HIV-infected Veterans and determine the relationship to health outcomes and care processes in these Veterans through review of medical records.

The investigators will use the VA medical record data, which allows for the study of the diverse VA patient population with patients from a range of personal backgrounds, geographic locations, and VA health care networks. HIV infection will be determined by the presence of two outpatient HIV diagnoses or one inpatient HIV diagnosis. This study will use a retrospective group of HIV-infected Veterans who used MHV between October 2007- October 2018 to evaluate the relationship between patient HIV care outcomes and MHV tool use. The investigators will look at data to carefully consider HIV-infected patient health status, health care received, and activity. The investigators will also look at Quality of Care (QC) outcomes which include medication adherence, CD4 count, viral load testing and detectable viral load, appointments, patient cancellations, patient no-shows, emergency department visits, flu vaccination, and syphilis and lipid testing. This aim/step will allow the investigators to examine differences in VA patients who have opted to use MHV versus those who have not opted to use MHV.

Aim/Step 2: Describe how Veterans with HIV use MHV for self-management, and why Veterans choose to use (or not to use) specific MHV tools; and similarly how and why providers use (or do not use) MHV.

The investigators will interview Veterans and providers to learn what motivates certain patients and providers/staff to use MHV in a certain way, or to understand MHV system issues, as well as attitudes and perceptions that prevent others from using MHV. The investigators will select patients and providers from six VA medical centers and interview those with high-, low, or no- MHV use. The investigators will discuss how participants use MHV to manage HIV and other conditions. The investigators will discuss with Veterans how providers use MHV as a tool for communication and coordination. With Veterans not using MHV (or minimal use), the investigators will ask about reasons. The interviews will be audio-recorded.

Aim/Step 3: Incorporate findings from Aims/Steps 1 and 2 to design an intervention that will be tested by Veterans and providers.

The investigators will compare the data from aims/steps 1 and 2 to develop an intervention that may improve self-management in Veterans with HIV. The investigators will identify Veterans and providers from two VA medical centers that will help the investigators test the intervention through "cognitive walkthroughs." Cognitive walkthroughs are used to test an intervention that is in the early stages of development. Veterans and providers will be the first to test if the intervention is acceptable and feasible. Participants will also offer feedback to the researchers as it relates to problems with using the intervention. The cognitive walkthroughs will be audio- and video-recorded.

Additional Aim a: Analyze qualitative data across the racial/ethnic and gender groups to evaluate MHV use, utilizing these findings to tailor interventions to racial/ethnic minority groups use an modified intervention mapping approach.

The investigators will develop an MHV intervention that meets the diversity of MHV user's needs, including Black and women Veterans. These findings could help MHV better understand how to target new interventions to potentially increase access to MHV and increase use of MHV for managing chronic conditions, among Black Veterans.

Additional Aim b: Develop a protocol for conducting virtual modified intervention mapping.

The investigators will develop the capability to conduct modified intervention mapping virtually. As no standard protocol has been developed for conducting intervention mapping virtually, the development of such protocol can contribute to lower cost, timely, and effective intervention design.

COVID-19 Expansion Aim 1: Explore historical trends of HIV clinical outcomes and indicators of care and trends observed during the COVID-19 pandemic, among Veterans living with HIV.

The investigators will use VA medical record data to examine these differences across racial/ethnic subgroups.

COVID-19 Expansion Aim 2: Use interrupted time series models to statistically compare pre-COVID-19 and COVID-19 pandemic HIV clinical outcomes and indicators of care.

The investigators will evaluate changes in disparities by expanding interrupted time series models to stratify by race/ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis (determined by the presence of two outpatient HIV diagnoses or one inpatient HIV diagnosis from 10/2007 to 10/2018)

Exclusion Criteria:

* Children under the age of 18
* Non-English speakers
* Those considered incompetent (as determined by the presence of an ICD-9/10 code for dementia or Alzheimer's)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consists of entire patient population of HIV-infected Veterans active in care at a VA Health Care System who are non-users of MHV or have used MHV.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Medical Record Review | 1 year
  Determine the relationship between MHV tools and quality of care and outcomes for Veterans who are HIV positive.
Interviews | 1 year
  Understand how Veterans with HIV use or choose not to use MHV for self-management
Intervention | 1 year
  Develop and test an intervention that will encourage use of MHV

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M. Midboe, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (8):
- United States (8):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Southern Nevada Healthcare System, North Las Vegas, NV, Las Vegas, Nevada
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Javier SJ, Troszak LK, Shimada SL, McInnes DK, Ohl ME, Avoundjian T, Erhardt TA, Midboe AM. Racial and ethnic disparities in use of a personal health record by veterans living with HIV. J Am Med Inform Assoc. 2019 Aug 1;26(8-9):696-702. doi: 10.1093/jamia/ocz024. PMID 30924875
- [Result] Giannitrapani KF, Fereydooni S, Silveira MJ, Azarfar A, Glassman PA, Midboe A, Zenoni M, Becker WC, Lorenz KA. How Patients and Providers Weigh the Risks and Benefits of Long-Term Opioid Therapy for Cancer Pain. JCO Oncol Pract. 2021 Jul;17(7):e1038-e1047. doi: 10.1200/OP.20.00679. Epub 2021 Feb 3. PMID 33534632
- [Result] Avoundjian T, Troszak L, Cave S, Shimada S, McInnes K, Midboe AM. Correlates of personal health record registration and utilization among veterans with HIV. JAMIA Open. 2021 Jun 16;4(2):ooab029. doi: 10.1093/jamiaopen/ooab029. eCollection 2021 Apr. PMID 34278241
- [Result] Conti J, Fix GM, Javier SJ, Cheng H, Perez T, Dunlap S, McInnes DK, Midboe AM. Patient and provider perspectives of personal health record use: a multisite qualitative study in HIV care settings. Transl Behav Med. 2023 Jul 1;13(7):475-485. doi: 10.1093/tbm/ibac118. PMID 37084300
- [Result] Midboe AM, Cave S, Shimada SL, Griffin AC, Avoundjian T, Asch SM, Gifford AL, McInnes DK, Troszak LK. Relationship Between Patient Portal Tool Use and Medication Adherence and Viral Load Among Patients Living with HIV. J Gen Intern Med. 2024 Feb;39(Suppl 1):127-135. doi: 10.1007/s11606-023-08474-z. Epub 2024 Jan 22. PMID 38252241